CLINICAL TRIAL: NCT06718530
Title: Characterization of Immune Genotypes and Antibody Profiles to Foster the discoVERY of diagnosticbioMARKERS of Liver Cancer Development
Acronym: VERYMARKERS
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2024-42
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatitis C virus (HCV), which infects more than 185 million people, is a major risk factor. Direct-acting antiviral (DAA) therapy has significantly improved the eradication of the virus, but has not completely eliminated the risk of HCC, so careful surveillance is necessary. The genetic diversity of the natural killer receptor, histocompatibility antigens (HLA) and interferon lambda 4 (INFL4) activity, among other factors, have been found to be crucial in directing disease progression. Importantly, these markers are detectable years before the diagnosis of HCC. In addition, polymorphic variants attributable to the expression of genes involved in innate-type immune response, such as IFNL4 and HLA-E, have been shown to be predictive for the development of HCC and have not yet been extensively studied. The aim of the study is to evaluate novel circulating biomarkers, including the presence of antibodies to specific HCV proteome peptides, IFNL4 expression, and the interaction of specific HLA receptors/ligands in a large cohort of HCV-positive subjects in order to create a screening strategy for the early diagnosis of HCV-associated HCC.

Part of the study will be devoted to describing the immune microenvironment associated with the expression of IFNL4 and HLAE, evaluating them as potential prognostic indicators for HCC in HCV-infected subjects undergoing surgery for HCC, as well as in those with advanced/metastatic HCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years with the presence of chronic infection, fibrosis, cirrhosis or HCV- associated HCC
* Patients able to understand and willing to sign the of informed consent
* Patients to answer the questions in the questionnaire of enrollment

Exclusion Criteria:

* Treatment for other oncological diseases
* Immunodepression congenital or acquired (HIV, organ transplantation, pharmacological)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with varying degrees of liver damage, diagnosed with of HCC or HCV-positive with diagnosed cirrhosis, fibrosis or long-term HCV infection
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in antibody profile between subjects with and without chronic HCV infection | up to 2 years
  Mean or median difference between the groups, as appropriate, will be calculated
Difference in antibody profile between subjects with chronic HCV infection receiving or not receiving DAA therapy | up to 2 years
  Mean or median difference between the groups, as appropriate, will be calculated

SECONDARY OUTCOMES:
Define a relationship between IgG levels toward HCV-specific peptides and viral load/development clinical after 2 years of follow-up | up to 2 years
  Correlation coefficient between the highest IgG levels towards at least one specific HCV peptide and high viral load will be calculated
Define a relationship between IgG levels toward HCV-specific peptides and HCV genotype | up to 2 years
  Relation will be analyzed with logistic regression analysis and represented with Odds Ratio (OR) and relative 95% Confidence Interval (95% CI)
Characterization of Interferon Lambda 4 (INFL4) and Human Leukocyte antigene (HLA-E) variants within patient with or without HCV related hepatocarcinoma (HCC) | up to 2 years
  Frequencies of genetic variants within patient with or without HCV related hepatocarcinoma (HCC) will be reported
Characterization of INFL4 and HLA-E variants within patient with or without HCV related chronic hepatitis | up to 2 years
  Frequencies of genetic variants within patient with or without HCV related chronic hepatitis will be reported
Define the mRNA pathways activated in the subjects with expression of INFL4 and of HLA-E | up to 2 years
  Data will be illustrated with volcano plot and heat map

CONTACTS AND LOCATIONS:
Overall Officials: Valli De Re, PhD, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO) - IRCCS; Renato Cannizzaro, MD, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO) - IRCCS
Locations (4):
- Italy (4):
  - Centro di Riferimento Oncologico (CRO) di aviano-IRCCS, Aviano, Pordenone
  - AORN S.Anna e S. Sebastiano, Via F. Palasciano, Caserta
  - Istituto Nazionale Tumori di Napoli, IRCCS "G. Pascale", Napoli
  - Dip. Univ. Clin. di Scienze mediche, chirurgiche e della salute Università di Trieste, Trieste